CLINICAL TRIAL: NCT05863234
Title: Multicenter, Open-label, Dose-escalation Phase I/II Study to Evaluate the Tolerability, Safety, Efficacy and Pharmacokinetics of Repeated Continuous Intravenous PPMX-T003 in Patients With Aggressive NK Cell Leukaemia (ANKL) (Physician-initiated Clinical Trial)
Brief Title: Safety Evaluation Study for Patients With Aggressive NK-cell Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hiroshima University Hospital (Other)
Collaborators: Kyoto University Hospital (Other); Hokkaido University Hospital (Other); Okayama University (Other); Tokai University (Other); Kyushu University (Other); Tohoku University (Other); Nagoya University (Other); Komagome Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPMX-T003-CT103
Record Dates: First submitted 2023-05-09; First posted 2023-05-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Aggressive NK Cell Leukemia
Keywords: neoplasms
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with PPMX-T003 (Experimental)
  Interventions: Drug: PPMX-T003

INTERVENTIONS:
Drug: PPMX-T003 — The therapeutic agent is administered continuously intravenously

SUMMARY:
This is Phase I/II Dose-Escalation Study to evaluate the tolerability, safety, efficacy and pharmacokinetics of PPMX-T003 in aggressive NK-cell leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ANKL (regardless of whether the disease is first or recurrent) based on diagnostic criteria developed with reference to the World Health Organization (WHO) 4th edition (2017) criteria.

Exclusion Criteria:

* Patients eligible to receive chemotherapy as treatment for ANKL

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of incidence of AEs and DLTs by PPMX-T003 repeated continuous intravenous administration (the first course) | 7days after the administration
  In order to evaluate tolerability and safety of PPMX-T003 repeated continuous intravenous administration in the first course, incidence of AEs and DLTs by the treatment are measured.

SECONDARY OUTCOMES:
Number of incidence of AEs and DLTs by PPMX-T003 repeated continuous intravenous administration (the second course or later) | From the second course to the final course (Max. 35days after the first administration)
  In order to evaluate tolerability and safety of PPMX-T003 repeated continuous intravenous administration in the second course or later, incidence of AEs and DLTs by the treatment are measured.
Efficacy of PPMX-T003 repeated continuous intravenous administration (1) Liver volume evaluated by CT scan | 35 days
  As a part of efficacy evaluation of the treatment, percentage change in the product of the maximum long and short diameters of the liver measured by CT (assessed by the primary physician)
Efficacy of PPMX-T003 repeated continuous intravenous administration (2) improvement in liver function as assessed by the Model for End-stage Liver Disease (MELD and MELD-Na) | 35 days
Efficacy of PPMX-T003 repeated continuous intravenous administration (3) Survival duration at 6 months | 6 months
Efficacy of PPMX-T003 repeated continuous intravenous administration (4) Percentage of subjects who were able to transition to chemotherapy | 35days after the treatment
Serum drug concentration during repeated continuous intravenous PPMX-T003 administration | 35 days
Anti-drug antibody production (Immunogenicity) | 35 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hiroshima University Hospital, Hiroshima, Hiroshima, Japan

REFERENCES:
- [Derived] Fukuhara N, Onizuka M, Kanda J, Asada N, Kato K, Ando K. Protocol for a multicentre, open-label, dose-escalation phase I/II study evaluating the tolerability, safety, efficacy and pharmacokinetics of repeated continuous intravenous PPMX-T003 in patients with aggressive natural killer cell leukaemia. BMJ Open. 2025 Jun 30;15(6):e098532. doi: 10.1136/bmjopen-2024-098532. PMID 40588385